CLINICAL TRIAL: NCT01219868
Title: Impact of Physician-nurse Team on ED Length of Stay
Brief Title: Physician-nurse Team to Reduce Emergency Department (ED) Overcrowding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Olivier T. Rutschmann, MD, MPH, University Hospital, Geneva
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SU-001
Record Dates: First submitted 2010-10-06; First posted 2010-10-13 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Triage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physician-nurse team (Experimental)
  Interventions: Behavioral: Physician-nurse team supervision

INTERVENTIONS:
Behavioral: Physician-nurse team supervision — Physician-nurse team will supervise patient's flow in the ED
  Other Names: No name

SUMMARY:
The objective of this study is to explore the impact of a physician-nurse team supervising patient's flow on ED length of stay

DETAILED DESCRIPTION:
A physician-nurse team will be in charge of patients flow in the ED during intervention periods. During control periods, no team will be present. The impact of this team on Ed length of stay will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients > 16 years presenting to the ED

Exclusion Criteria:

* no

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8000 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
ED length of stay | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier T Rutschmann, MD, MPH, Principal Investigator — HUG
Locations (1):
- ED of Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland